CLINICAL TRIAL: NCT00028431
Title: An Open Label Study of MDX-CTLA4 in Combination With Tyrosinase/gp100/MART-1 Peptides Emulsified With Montanide ISA 51 in the Treatment of Patients With Resected Stage III or IV Melanoma
Brief Title: Novel Adjuvants for Peptide-Based Melanoma Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-R-1975-01; 10M-00-4;; FD-R-001975-01
Record Dates: First submitted 2002-01-04; First posted 2002-01-09 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma
Keywords: Stage III melanoma; Stage IV melanoma; Interleukin-12; Cancer Vaccines; Antineoplastic Agents, Combined; Incomplete Freund's adjuvant; Monophenol Monooxygenase; Mannitol; Adjuvants, Immunologic; Melan-A Protein; Antigens, Neoplasm; Antibodies; Melanocyte lineage-specific antigen gp100; CTLA-4
MeSH Terms: conditions — Melanoma; Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Monophenol Monooxygenase

INTERVENTIONS:
Biological: MDX-CTLA4 Antibody; Tyrosinase/gp100/MART-1 Peptides Melanoma Vaccine

SUMMARY:
This is a study to determine the efficacy of a melanoma vaccine chemotherapy cocktail composed of CTLA-4 antibody; tyrosinase, gp100, and MART-1 peptides; and incomplete Freund's adjuvant (IFA) with or without interleukin-12 in patients with resected stage III or IV melanoma.

DETAILED DESCRIPTION:
In the Phase I/II trial, patients with resected stages III and IV melanoma who have been rendered free of disease, but are at high risk of relapse, are treated with peptides/IFA at a dose of 0.5 mg each peptide plus CTLA-4 antibody given intravenously, 3 mg/kg, after each vaccination. In the Phase II randomized study, patients are treated with the melanoma peptide vaccine alone, with CTLA-4 antibody, or with CTLA-4 antibody combined with IL-12 at 30 ng/kg with alum. The peptides are tyrosinase 368-376 (370D); gp100 209-217 (210M); and MART-1 26-35 (27L) which are emulsified with IFA. The dosing schedule for both trials are at 1, 2, 3, 4, 5, and 6 months; then at 9 and 12 for a total of 8 vaccinations.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of stage III or IV cutaneous, mucosal, or ocular melanoma
* Completely resected disease or disease-free
* HLA-A2.1 positive
* Tumor tissue available for immunohistochemical analysis and staining positive for at least 1 of the specified antigens
* At least 1 month since prior therapy for cancer, including radiotherapy and adjuvant therapy
* WBC count at least 3,000/mm3
* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9.0 gm/dL
* Creatinine no greater than 2.0 mg/dL
* Bilirubin no greater than 2.0 mg/dL
* SGOT/SGPT no greater than 2.5 times upper limit of normal
* ECOG performance status 0-1
* Have failed alpha-interferons (patients with resected stage III disease)

Exclusion criteria:

* Prior treatment with tyrosinase: 368-376(370D), gp100:209-217(210M), and MART-1:26-35(27L) peptides
* Steroid therapy or other immunosuppressive medication requirement
* Major systemic infections (e.g., pneumonia or sepsis)
* Coagulation or bleeding disorders
* Major medical illnesses of the gastrointestinal, cardiovascular, or respiratory systems
* Allergic reaction to Montanide ISA 51 (incomplete Freund's adjuvant)
* History of uveitis or autoimmune inflammatory eye disease
* Other active autoimmune disease
* Positive for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-08; Primary Completion 2003-01 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, M.D., Ph.D., Principal Investigator — University of Southern California/Norris Cancer Center
Locations (1):
- Universtiy of Southern California/Kenneth Norris, Jr. Comprehensive Cancer Center, Los Angeles, California, United States